CLINICAL TRIAL: NCT02761512
Title: A Double Blind, Randomized, Active-controlled, Phase 3 Study to Evaluate the Safety and Efficacy of CJ-12420 in Patients With Gastric Ulcer
Brief Title: Study to Evaluate the Safety and Efficacy of CJ-12420 in Patients With Gastric Ulcer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: HK inno.N Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CJ_APA_303
Record Dates: First submitted 2016-05-01; First posted 2016-05-04 (Estimated); Last update posted 2019-08-22 (Actual); Status verified 2018-04

CONDITIONS: Gastric Ulcer
MeSH Terms: conditions — Stomach Ulcer | interventions — Lansoprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- CJ-12420 50 mg QD (Experimental): CJ-12420 50 mg, tablet, once daily, oral administration for up to 8 weeks
  Interventions: Drug: CJ-12420 50 mg QD
- CJ-12420 100 mg QD (Experimental): CJ-12420 100 mg, tablet, once daily, oral administration for up to 8 weeks
  Interventions: Drug: CJ-12420 100 mg QD
- Lansoprazole 30 mg QD (Active Comparator): Lansoprazole 30 mg, capsule, once daily, oral administration for up to 8 weeks
  Interventions: Drug: Lansoprazole 30 mg QD

INTERVENTIONS:
Drug: CJ-12420 50 mg QD — CJ-12420 50 mg tablets will be orally administered, once daily, for up to 8 weeks. For subjects whose gastric ulcer is not endoscopically healed(S1 or S2 stage) at Week 4, subjects will receive additional 4 weeks treatment of CJ-12420 50 mg.
  Other Names: Not yet decided
  Arms: CJ-12420 50 mg QD
Drug: CJ-12420 100 mg QD — CJ-12420 100 mg tablets will be orally administered, once daily, for up to 8 weeks. For subjects whose gastric ulcer is not endoscopically healed(S1 or S2 stage) at Week 4, subjects will receive additional 4 weeks treatment of CJ-12420 100 mg.
  Other Names: Not yet decided
  Arms: CJ-12420 100 mg QD
Drug: Lansoprazole 30 mg QD — Lansoprazole 30 mg capsule will be orally administered, once daily, for up to 8 weeks. For subjects whose gastric ulcer is not endoscopically healed(S1 or S2 stage) at Week 4, subjects will receive additional 4 weeks treatment of Lansoprazole 30 mg.
  Other Names: Lanston cap.
  Arms: Lansoprazole 30 mg QD

SUMMARY:
To demonstrate non-inferiority of CJ-12420 to lansoprazole 30 mg capsule in terms of therapeutic efficacy, and to confirm safety of CJ-12420, after once daily oral administration of CJ-12420 50 mg, 100 mg or Lansoprazole 30 mg capsule in gastric ulcer patients.

DETAILED DESCRIPTION:
This is a double blind, randomized, placebo-controlled, phase 3 study. Subjects will be randomly assigned to one of the three treatment groups (CJ-12420 50 mg, 100 mg or Lansoprazole 30 mg).

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of 1 or more active gastric ulcers (≥3 mm ~ ≤30 mm using open biopsy forceps) according to the Sakita-Miwa classification (A1 or A2 stage) from upper GI endoscopy at the same institution within 14 days prior to initiation of the investigational product administration.

Exclusion Criteria:

1. Finding of gastrointestinal bleeding, esophageal stricture, ulcer stenosis, pyloric stenosis, esophageal gastric varices, Barrett's esophageal of >3 cm (long segment Barrett esophagus, LSBE), duodenal ulcer, intractable ulcer, digestive ulcer perforation or malignancy on upper GI endoscopy.
2. Ulcer caused by an endoscopic surgery (e.g., ulcer after EMR/ESD)
3. Requirement of persistent daily use of drugs that may cause an ulcer such as nonsteroidal anti-inflammatory drugs(NSAIDs) or aspirin during the course of the study
4. Scheduled surgery requiring hospitalization or requirement of surgical treatment during study participation
5. Subjects who participated in the other clinical trial within 4 weeks prior to randomization

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 306 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2018-07-26 (Actual); Study Completion 2018-12-28 (Actual)

PRIMARY OUTCOMES:
Cumulative healing rate of gastric ulcer at 8-week | 8 weeks

SECONDARY OUTCOMES:
Healing rate of gastric ulcer at 4-week | 4 weeks
Week 8 healing rates by H. pylori infection | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Myung Gyu Choi, M.D., Ph.D, Principal Investigator — Catholic Univ. Seoul St. Mary Hospital
Locations (2):
- South Korea (2):
  - Catholic Univ. Seoul St. Mary Hospita, Seoul
  - Kyung Hee University Medical Center, Seoul

IPD SHARING:
Plan to Share IPD: No